CLINICAL TRIAL: NCT05666115
Title: Efficacy of Modification of Lifestyle in the Treatment of Ankylosing Spondylitis
Brief Title: Efficacy of Modification of Lifestyle in the Treatment of Ankylosing Spondylitis: a Pilot Study
Acronym: EMLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Elena Sonsoles Rodriguez López, Principal Investigator, Camilo Jose Cela University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMLAS
Record Dates: First submitted 2022-11-22; First posted 2022-12-27 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Arthritis; Rheumatic Diseases; Autoimmune Diseases
MeSH Terms: conditions — Arthritis; Rheumatic Diseases; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Participants in the probiotics group will receive probiotic supplementation for 12 weeks.
  Interventions: Dietary Supplement: Probiotic group
- Exercise group (Active Comparator): The control group will undergo a 12-week online-delivered Tabata program, as a form of high-intensity interval training.
  Interventions: Other: Exercise group

INTERVENTIONS:
Dietary Supplement: Probiotic group — During the first 4 weeks, patients will be instructed to take two capsules of Enterelle plus (Bromatech lab, Manno, Switzerland) during morning time, before or after breakfast. Enterelle plus contains specific strains, i.e., S boulardi, E faecium, and acidophilus, that contribute to reduce the mycotic flora and modulate the gastrointestinal transit. For the next 8 weeks, participants will be told to ingest two capsules of Adomelle (Bromatech lab, Manno, Switzerland) at night, during or right after dinner. Adomelle contains several strains, including Bifidobacterium breve, that help to reduce abdominal fat, pain, and gas, and control the frequency of deposition
  Arms: Probiotic group
Other: Exercise group — This type of intervention has shown to benefit patients with several chronic conditions 23, including axSpA 13. Exercises combined high knees, lunges, basic burpees, plank, skipping, mountain climbers, and squats with jumps. The training routine will be conducted three times per week, and each session will last around 8 minutes (2 sets of 4 minutes, with a 10 second rest between them). All sessions will be individually tailored and supervised by a senior professional with a degree in Physiotherapy and Sciences of Physical Activity and Sport. Overall, participants will be told to continue exercising if low to moderate bearable pain appeared during training.
  Arms: Exercise group

SUMMARY:
Axial spondyloarthritis (axSpA) is a chronic inflammatory immune disorder with a global prevalence that ranges from 20 to 160 cases per 10000 individuals. axSpA has two forms of clinical presentation (radiographic and non-radiographic) based on the presence or absence of radiographic sacroiliitis. This condition mostly affects the vertebral spine, and is characterized by joint pain and stiffness, fatigue, and restricted function, which leads to a substantial physical, psychological, and socioeconomic burden. The clinical management of axSpA needs to combine pharmacological and non-pharmacological approaches to reduce inflammation and improve health-related quality of life.

The aim of the study will be to determine if a 12-week probiotic supplementation will be more effective than an online-delivered strength training program at improving functional capacity in adults with non-radiographic axSpA. As a secondary aim, we will compare the impact of both interventions on disease activity, spinal mobility, quality of life and biochemical measures. This will be the first randomized controlled trial where probiotics are compared with an active intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18 years or older and have a confirmed diagnosis of non-radiographic axSpA following the 2009 Assessment of the SpondyloArthritis International Society classification criteria

Exclusion Criteria:

* Any systemic disease or comorbidity that may severely impair exercise capacity.
* A high sensitivity C-reactive protein 10-fold greater than the normal upper limit (2.87 mg/l).
* Any changes to medical treatment within the previous 2 months, and having an active peripheral arthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be functional disability during daily life activities, evaluated with the Bath Ankylosing Spondylitis Functional Index. | Change from Baseline BASFI at 4 and 12 weeks
  The Bath Ankylosing Spondylitis Functional Index includes 10 items (scale of 0 to 10, higher scores denoting worse performance), and is among the recommended core set of instruments for axSpA.

SECONDARY OUTCOMES:
The secondary outcome will be disease activity during daily life activities, evaluated with the Bath Ankylosing Spondylitis Disease Activity Index. | Change from Baseline BASDAI at 4 and 12 weeks
  Disease activity will be assessed with the Bath Ankylosing Spondylitis Disease Activity Index. The Bath Ankylosing Spondylitis Disease Activity Index explores five different constructs (fatigue, spinal or peripheral joint pain, localized tenderness, and morning stiffness), with lower scores representing less disease activity (scale of 0 to 10).
Spinal mobility will be measured with the Bath Ankylosing Spondylitis Metrology Index (BASMI) | Change from Baseline BASMI at 4 and 12 weeks
  Bath Ankylosing Spondylitis Metrology Index as a composite index including lumbar flexion and side flexion (cm), tragus-to-wall and intermalleolar distance (cm), and cervical rotation (degrees). Final scores of the BASMI range from 0 "no mobility limitation" to 10 "severe limitation".
The Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) 30 will be used to determine health-related quality of life | Change from Baseline ASQoL at 4 and 12 weeks
  The ASQoL is valid, feasible and reliable. Total score range between 0 and 18, with higher scores indicating poorer quality of life.
Biochemical measures (interleukin-1 (IL-1) and tumor necrosis factor a (TNFa)) | Change from Baseline biochemical measures at 4 and 12 weeks
  A PeliKine compact enzyme-linked immunosorbent assay (ELISA) kit will be used to explore two inflammatory biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Sonsoles Rodriguez Lopez, Arroyomolinos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No